CLINICAL TRIAL: NCT00148733
Title: Community- and Health Facility-based Intervention With Zinc as Adjuvant Therapy for Pneumonia to Enhance Child Health and Nutrition
Brief Title: CHIZAP: Community- and Health Facility-Based Intervention With Zinc as Adjuvant Therapy for Childhood Pneumonia
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Centre For International Health (Other)
Collaborators: Tribhuvan University, Nepal (Other); Statens Serum Institut (Other); All India Institute of Medical Sciences (Other); IRD, Epidemiologie et Prevention, Montpelier, France (Unknown); Society for Applied Studies (Other)
Responsible Party: Principal Investigator, Tor A. Strand, Professor, Centre For International Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 003740; 003740(Eur. Comm. INCO) (Other Grant/Funding Number: European Union); NUFU PRO 36/2002 (Other Grant/Funding Number: NUFU)
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Results first posted 2015-02-16 (Estimated); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Pneumonia
Keywords: Child; pneumonia; Zinc; clinical trial; Nepal; nutrition; therapeutic
MeSH Terms: conditions — Pneumonia | interventions — Zinc

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Zinc (Experimental): Zinc sulphate 10 or 20 mg (elemental zinc) per day. Intervention and placebo given perorally mixed with approximately 5 mL of breastmilk or clean water
  Interventions: Drug: Zinc
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Zinc

INTERVENTIONS:
Drug: Zinc — Dissolvable zinc tablet 10 mg elemental zinc per day for infants 20 mg elemental zinc per day for children 12 to 35 months
  Other Names: Produced by Nutriset, Malaunay, France

SUMMARY:
The aim of the study described is to measure the degree with which zinc given as adjunct therapy to standard antibiotic treatment during childhood pneumonia reduces the risk of treatment failure and the duration of the illness.

DETAILED DESCRIPTION:
Hypothesis: Zinc deficiency is a major public health problem in developing counties. Poor zinc status is associated with stunted growth and reduced resistance to infections. Several in vitro experiments and in vivo studies in animals and humans have demonstrated detrimental effects of zinc depletion on almost all facets of the immune system. The epithelial linings in the gut and in the respiratory tract are important for the resistance to infections and continuous cell division is required for proper function of these barriers. Zinc is crucial for cellular division and for the maintenance of organs with cells with a rapid turnover, including epithelial cells. Clinical trials in children in developing countries have demonstrated improved growth and reduced prevalence of diarrhea and respiratory tract infections following zinc supplementation. Furthermore, zinc has a well-documented therapeutic effect when given during acute or persistent diarrhea. The effect of zinc may be explained by correction of a deficiency state and/or by a pharmacological, as yet poorly described, action.

Due to the promising results from previous studies, WHO are now supporting large clinical trials in Nepal, India and Tanzania to assess whether routine zinc supplementation reduces mortality in early childhood. If the results of these trials show a mortality reduction, routine zinc supplementation or zinc dense foods may be promoted. However, while the first approach is logistically difficult and expensive, the second approach is difficult because zinc dense foods and foods with low phytic acid content are expensive and not readily available. Moreover, both approaches may be perceived to be incompatible with the current breast-feeding recommendations for the youngest children in most developing countries.

There is limited information on zinc as adjunct therapy for pneumonia. A recent hospital-based study in young children with severe pneumonia, showed that the zinc group had a faster recovery, resulting in a shortening of stay in hospital of one day. However, this study was small and no community based study has been conducted so far. Whether zinc has an effect during respiratory infections has to be assessed in studies with larger sample sizes in children with less severe disease and should be repeated in children with more severe disease. Short-term zinc administration during infections may become an alternative or an addition to long-term supplementation or promotion of zinc dense foods. Furthermore, therapeutic administration of zinc will not interfere with the current breast-feeding recommendations.

Hypothesis: Zinc as adjunct therapy for pneumonia may lead to faster recovery. Furthermore, long-term beneficial effects may include improved immuno-nutritional status measured by thymus size, less morbidity and improved growth.

Comparison: Duration of illness, risk of treatment failure, for those with severe pneumonia: length of hospital stay. Number of non-injury clinic visits and hospitalizations during the intervention with Zinc and an in a 6 month period after enrolment. Growth assessed by anthropometry and thymus size assessed by ultrasonography. Explore the efficacy of zinc in etiology-sub groups including those defined by nutritional status, inflammation, fever, gender, breastfeeding status and viral etiology.

ELIGIBILITY:
Inclusion Criteria:

* Pneumonia: Child presenting with cough or difficult breathing and elevated respiratory rate.
* Severe pneumonia: Child presenting with cough or difficult breathing and chest indrawing , but without any of the following danger signs:

  * not able to drink/breastfeed,
  * vomit everything,
  * has had convulsions,
  * is lethargic or unconscious.
* Must be able to take Zinc

Exclusion Criteria:

* The child requires special care for severe illness other than pneumonia
* Severe malnutrition defined as being < 70% National Center for Health Statistics (NCHS) median weight for height
* Presence of congenital heart disease
* Documented tuberculosis
* Any antibiotic treatment during the last 48 hours
* The child was enrolled less than 6 months ago
* Presence of dysentery
* Cough for more than 14 days

Ages: 2 Months to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2628 (Actual)
Dates: Start 2004-01; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tor A Strand, MD PhD, Principal Investigator — Centre for International Health, University of Bergen, 5021 Bergen, Norway; Halvor Sommerfelt, MD PhD, Study Director — Centre for International Health, University of Bergen, 5021 Bergen, Norway; Prakash S Shrestha, MD Professor, Study Director — Child Health Research Project, Department of Child Health, Institute of Medicine, Maharajganj; Ramesh K Adhikari, MD Dean, Study Chair — Child Health Research Project, Department of Child Health, Institute of Medicine, Maharajganj; Palle Valentiner-Branth, MD PhD, Principal Investigator — Department of Epidemiology Research, Statens Serum Institut, 2300 Copenhagen S, Denmark
Locations (1):
- Siddhi Memorial Hospital (SMH),Bhelukhel, Bhimsensthan, Bhaktapur, Nepal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bhutta ZA, Black RE, Brown KH, Gardner JM, Gore S, Hidayat A, Khatun F, Martorell R, Ninh NX, Penny ME, Rosado JL, Roy SK, Ruel M, Sazawal S, Shankar A. Prevention of diarrhea and pneumonia by zinc supplementation in children in developing countries: pooled analysis of randomized controlled trials. Zinc Investigators' Collaborative Group. J Pediatr. 1999 Dec;135(6):689-97. doi: 10.1016/s0022-3476(99)70086-7. PMID 10586170
- [Background] Bates CJ, Prentice A. Breast milk as a source of vitamins, essential minerals and trace elements. Pharmacol Ther. 1994 Apr-May;62(1-2):193-220. doi: 10.1016/0163-7258(94)90011-6. PMID 7991643
- [Background] Walsh CT, Sandstead HH, Prasad AS, Newberne PM, Fraker PJ. Zinc: health effects and research priorities for the 1990s. Environ Health Perspect. 1994 Jun;102 Suppl 2(Suppl 2):5-46. doi: 10.1289/ehp.941025. PMID 7925188
- [Background] Strand TA, Chandyo RK, Bahl R, Sharma PR, Adhikari RK, Bhandari N, Ulvik RJ, Molbak K, Bhan MK, Sommerfelt H. Effectiveness and efficacy of zinc for the treatment of acute diarrhea in young children. Pediatrics. 2002 May;109(5):898-903. doi: 10.1542/peds.109.5.898. PMID 11986453
- [Background] Bates CJ, Evans PH, Dardenne M, Prentice A, Lunn PG, Northrop-Clewes CA, Hoare S, Cole TJ, Horan SJ, Longman SC, et al. A trial of zinc supplementation in young rural Gambian children. Br J Nutr. 1993 Jan;69(1):243-55. doi: 10.1079/bjn19930026. PMID 8457531
- [Background] Black RE. Therapeutic and preventive effects of zinc on serious childhood infectious diseases in developing countries. Am J Clin Nutr. 1998 Aug;68(2 Suppl):476S-479S. doi: 10.1093/ajcn/68.2.476S. PMID 9701163
- [Background] Sazawal S, Black RE, Jalla S, Mazumdar S, Sinha A, Bhan MK. Zinc supplementation reduces the incidence of acute lower respiratory infections in infants and preschool children: a double-blind, controlled trial. Pediatrics. 1998 Jul;102(1 Pt 1):1-5. doi: 10.1542/peds.102.1.1. PMID 9651405
- [Background] Bhandari N, Bahl R, Taneja S, Strand T, Molbak K, Ulvik RJ, Sommerfelt H, Bhan MK. Effect of routine zinc supplementation on pneumonia in children aged 6 months to 3 years: randomised controlled trial in an urban slum. BMJ. 2002 Jun 8;324(7350):1358. doi: 10.1136/bmj.324.7350.1358. PMID 12052800
- [Background] Hambidge KM, Krebs NF, Miller L. Evaluation of zinc metabolism with use of stable-isotope techniques: implications for the assessment of zinc status. Am J Clin Nutr. 1998 Aug;68(2 Suppl):410S-413S. doi: 10.1093/ajcn/68.2.410S. PMID 9701153
- [Background] Chai F, Truong-Tran AQ, Ho LH, Zalewski PD. Regulation of caspase activation and apoptosis by cellular zinc fluxes and zinc deprivation: A review. Immunol Cell Biol. 1999 Jun;77(3):272-8. doi: 10.1046/j.1440-1711.1999.00825.x. PMID 10361260
- [Background] Truong-Tran AQ, Carter J, Ruffin R, Zalewski PD. New insights into the role of zinc in the respiratory epithelium. Immunol Cell Biol. 2001 Apr;79(2):170-7. doi: 10.1046/j.1440-1711.2001.00986.x. PMID 11264713
- [Background] Shankar AH, Prasad AS. Zinc and immune function: the biological basis of altered resistance to infection. Am J Clin Nutr. 1998 Aug;68(2 Suppl):447S-463S. doi: 10.1093/ajcn/68.2.447S. PMID 9701160
- [Background] Lira PI, Ashworth A, Morris SS. Effect of zinc supplementation on the morbidity, immune function, and growth of low-birth-weight, full-term infants in northeast Brazil. Am J Clin Nutr. 1998 Aug;68(2 Suppl):418S-424S. doi: 10.1093/ajcn/68.2.418S. PMID 9701155
- [Background] Bhandari N, Bahl R, Taneja S, Strand T, Molbak K, Ulvik RJ, Sommerfelt H, Bhan MK. Substantial reduction in severe diarrheal morbidity by daily zinc supplementation in young north Indian children. Pediatrics. 2002 Jun;109(6):e86. doi: 10.1542/peds.109.6.e86. PMID 12042580
- [Background] Brooks WA, Yunus M, Santosham M, Wahed MA, Nahar K, Yeasmin S, Black RE. Zinc for severe pneumonia in very young children: double-blind placebo-controlled trial. Lancet. 2004 May 22;363(9422):1683-8. doi: 10.1016/S0140-6736(04)16252-1. PMID 15158629
- [Background] Bhandari N, Bahl R, Hambidge KM, Bhan MK. Increased diarrhoeal and respiratory morbidity in association with zinc deficiency--a preliminary report. Acta Paediatr. 1996 Feb;85(2):148-50. doi: 10.1111/j.1651-2227.1996.tb13981.x. PMID 8640039
- [Background] Sazawal S, Black RE, Bhan MK, Jalla S, Sinha A, Bhandari N. Efficacy of zinc supplementation in reducing the incidence and prevalence of acute diarrhea--a community-based, double-blind, controlled trial. Am J Clin Nutr. 1997 Aug;66(2):413-8. doi: 10.1093/ajcn/66.2.413. PMID 9250122
- [Background] Sazawal S, Black RE, Bhan MK, Bhandari N, Sinha A, Jalla S. Zinc supplementation in young children with acute diarrhea in India. N Engl J Med. 1995 Sep 28;333(13):839-44. doi: 10.1056/NEJM199509283331304. PMID 7651474
- [Background] Integrated management of the sick child. Bull World Health Organ. 1995;73(6):735-40. PMID 8907767
- [Derived] Haugen J, Chandyo RK, Brokstad KA, Mathisen M, Ulak M, Basnet S, Valentiner-Branth P, Strand TA. Cytokine Concentrations in Plasma from Children with Severe and Non-Severe Community Acquired Pneumonia. PLoS One. 2015 Sep 25;10(9):e0138978. doi: 10.1371/journal.pone.0138978. eCollection 2015. PMID 26407163
- [Derived] Valentiner-Branth P, Shrestha PS, Chandyo RK, Mathisen M, Basnet S, Bhandari N, Adhikari RK, Sommerfelt H, Strand TA. A randomized controlled trial of the effect of zinc as adjuvant therapy in children 2-35 mo of age with severe or nonsevere pneumonia in Bhaktapur, Nepal. Am J Clin Nutr. 2010 Jun;91(6):1667-74. doi: 10.3945/ajcn.2009.28907. Epub 2010 Apr 7. PMID 20375190

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Zinc | Placebo
Started | 1314 | 1314
Completed | 1300 | 1299
Not Completed | 14 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Zinc | Placebo | Total
Number analyzed (Participants) | 1314 | 1314 | 2628
Age, Continuous [Mean (Standard Deviation); unit: months] | 7.3 (7.4) | 7.2 (7.2) | 7.2 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 575 | 576 | 1151
  Male | 739 | 738 | 1477

OUTCOME MEASURES:

1. Primary Outcome: Risk of Treatment Failure.
Description: Enrolled children will be followed and given zinc or placebo for 14 days. We will compare the proportion with treatment failure (i.e. lack of improvement within 3 days) between the two groups
Time Frame: Within 2 weeks after enrollment
Measure: Number; unit: participants
Arm/Group | Zinc | Placebo
Number analyzed (Participants) | 1300 | 1299
participants | 267 | 253

2. Primary Outcome: Non-injury Clinic Visits and Hospital Admissions After Treatment Has Been Initiated
Description: We will measure to what extent the intervention can reduce the number of severe events.
Time Frame: Within 2 weeks after enrollment
Reporting Status: Not Posted, anticipated posting 2024-12

3. Primary Outcome: Active and Passive Morbidity Surveillance for Six Months After the 14-day Supplementation Period is Completed
Description: We will measure to what extent short term zinc administration has an impact on growth and morbidity for up to 6 months after end of supplementation
Time Frame: six months
Reporting Status: Not Posted, anticipated posting 2024-12

4. Primary Outcome: Difference in Growth and Thymic Size Between the Treatment Groups Measured at Three and Six Months After the Zinc Supplementation
Description: Thymus size will be measured using ultrasonography and compared between the two groups. at two occasions 2.5 and 6 months after end of supplementation
Time Frame: six months
Reporting Status: Not Posted, anticipated posting 2024-12

5. Primary Outcome: Adverse Effects
Description: Vomiting, regurgitation, pain in abdomen for 15 minutes after zinc or placebo administration.
Time Frame: 14 days
Reporting Status: Not Posted, anticipated posting 2024-12

6. Secondary Outcome: Effect Modifiers for the Effect of Zinc Given During Pneumonia
Description: We will also measure of there are factors at baseline that modifies the effect of zinc. Whether the following are modifiers for the above-mentioned effect of zinc given during pneumonia: i.severe inflammation, reflected in: high fever and/or elevated plasma C-reactive protein (CRP) concentration
Time Frame: Within 2 weeks after enrollment
Reporting Status: Not Posted, anticipated posting 2024-12

7. Secondary Outcome: The Efficacy of Zinc According to Breast Feeding Status and in Different Age Categories
Description: We will measure to what extent breastfeeding status modifies the effect of zinc on pneumonia
Time Frame: Within 2 weeks after enrollment
Reporting Status: Not Posted, anticipated posting 2024-12

8. Secondary Outcome: The Efficacy of Zinc in Malnourished and Non-malnourished Children
Description: We will compare the efficacy of zinc in those that are stunted, wasted or underweight with those who are not.
Time Frame: Within 2 weeks after enrollment
Reporting Status: Not Posted, anticipated posting 2024-12

9. Secondary Outcome: Will Presence of a RNA Virus Modify the Effect of Zinc
Description: We will compare the efficacy of zinc according to virus detected in nasopharyngeal secretions
Time Frame: 14 days
Reporting Status: Not Posted, anticipated posting 2024-12

10. Secondary Outcome: Folate, Cobalamin and Vitamin D Status of the Enrolled Children
Description: And whether or not these vitamins predict treatment failure and duration of illness.
Time Frame: 14 days
Reporting Status: Not Posted, anticipated posting 2024-12

ADVERSE EVENTS:
Time Frame: 14 days, while zinc or placebo were given
Description: Vomiting following zinc or placebo supplementation
Arm/Group | Zinc | Placebo
Serious Adverse Events (participants affected / at risk) | 0/1314 | 0/1314
Other Adverse Events (participants affected / at risk) | 181/1314 | 53/1314
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Zinc (N=1314) | Placebo (N=1314)
Regurgitation (Gastrointestinal disorders) | 181 | 53 — Study staff were observing the participants for 30 minutes after each dose of zinc or placebo.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No